CLINICAL TRIAL: NCT02993172
Title: The Copenhagen City Heart Study 'Østerbroundersøgelsen'
Brief Title: The Copenhagen City Heart Study
Acronym: CCHS
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Eva Prescott, Professor, Bispebjerg Hospital
Other Study IDs: CCHS
Record Dates: First submitted 2016-12-09; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Heart Disease; Stroke; Heart Failure; Cancer; Myocardial Infarction; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Coronary Disease; Stroke; Heart Failure; Neoplasms; Myocardial Infarction; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Copenhagen City Heart Study is an ongoing cardiovascular population study initiated in 1976 which has examined approximately 25,000 individuals from the general population. The initial sample has been re-invited up to four times and supplemented by younger individuals. The study includes questionnaires, clinical assessment and biomarkers. The population have been followed in a number of outcome registries and more than 900 scientific papers have been published.

DETAILED DESCRIPTION:
The Copenhagen City Heart Study, also known as "Østerbroundersøgelsen", is a large prospective cardio-vascular population study of 20,000 women and men that was launched in 1975 by Dr Peter Schnohr and Dr Gorm Jensen together with statistician Jørgen Nyboe and Prof. A. Tybjærg Hansen.

The original purpose of the study was to focus on prevention of coronary heart disease and stroke. During the years many other aspects have been added to the study: pulmonary diseases, heart failure, arrhythmia, alcohol, arthrosis, eye diseases, allergy, epilepsia, dementia, stress, vital exhaustion, social network, sleep-apnoe, ageing and genetics. In the fourth and fifth wave of the examination echocardiography was included.

The Copenhagen City Heart Study has invited a random sample of the census population in an area of central Copenhagen in five waves. The primary population was a random sample of 19,329 men and women 20-93 years old, drawn from a population of approximately 90,000 inhabitants aged 20 years or older living in a central part of Copenhagen (Østerbro). Using the unique personal identification number (Central-Personal-Register-code), consisting of date of birth and a registration number, the sample was age-stratified within 5-year age groups, with the main emphasis on the age groups from 35 to 70 years. The total number of participants invited to the first four examinations was: 19,329+500+3,000+1,062 = 23,891 men and women. Of the original 14,223 examined at the first examination 3,092 (21.7%) have been examined in all four examinations.

Follow-up of mortality and morbidity using the unique personal identification number is performed by linkage to a number of nation-wide disease registries. Follow-up completion rate is almost 100 percent (less than 0.1% have been lost to follow-up mainly through emigration), which is very uncommon for large population studies.

Overview of the patients examined in the Copenhagen City Heart Study:

1. st exam: 1976-78, 19,329 invited, 14,223 (73.6%) attended
2. nd exam: 1981-83, 18,059 invited, 12,698 (71.2%) attended
3. rd exam: 1991-94, 16,563 invited, 10.135 (61.2%) attended
4. th exam: 2001-03,12,600 invited, 6,238 (49.5%) attended
5. th exam: 2011-2014, approx 10,000 invited, approx 5000 (50%) attended

The Copenhagen City Heart Study is governed by a Steering Committee. The data from the Copenhagen City Heart Study is made available to researchers upon application to and approval by the Steering Committee. The following constitute the Steering Committee:

Gorm Jensen and Peter Schnohr (initiators), Peter Lange, Eva Prescott, Børge Nordestgaard, Morten Grønbæk, Anne Tybjærg Hansen, Stig Bojesen, Finn Gyntelberg, Jan Skov Jensen and Merete Appleyard

ELIGIBILITY:
Inclusion Criteria:

* Background population living in a defined area of Copenhagen

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age.stratified random sample of the census population
Sampling Method: Non-Probability Sample
Enrollment: 23891 (Actual)
Dates: Start 1976-01; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Registry based disease outcomes, mainly cardiovascular, pulmonary and cancer outcomes | Latest registry update december 31 2014

REFERENCES:
- [Derived] Larsen BS, Olsen FJ, Andersen DM, Madsen CV, Mogelvang R, Jensen GB, Schnohr P, Aplin M, Host NB, Christensen H, Sajadieh A, Biering-Sorensen T. Left Atrial Volumes and Function, and Long-Term Incidence of Ischemic Stroke in the General Population. J Am Heart Assoc. 2022 Sep 20;11(18):e027031. doi: 10.1161/JAHA.122.027031. Epub 2022 Sep 8. PMID 36073645
- [Derived] Olsen FJ, Skaarup KG, Lassen MCH, Johansen ND, Sengelov M, Jensen GB, Schnohr P, Marott JL, Sogaard P, Gislason G, Svendsen JH, Mogelvang R, Aalen JM, Remme EW, Smiseth OA, Biering-Sorensen T. Normal Values for Myocardial Work Indices Derived From Pressure-Strain Loop Analyses: From the CCHS. Circ Cardiovasc Imaging. 2022 May;15(5):e013712. doi: 10.1161/CIRCIMAGING.121.013712. Epub 2022 May 10. PMID 35535593
- [Derived] Svendstrup M, Allin KH, Angquist L, Schnohr P, Jensen GB, Linneberg A, Thuesen B, Astrup A, Saris WHM, Vestergaard H, Sorensen TIA. Is abdominal obesity at baseline influencing weight changes in observational studies and during weight loss interventions? Am J Clin Nutr. 2018 Nov 1;108(5):913-921. doi: 10.1093/ajcn/nqy187. PMID 30475965